CLINICAL TRIAL: NCT02375789
Title: Intranasal Evaporative COOLing for the Symptomatic Relief of Migraine HEADache - A Randomized, Double Blind, Placebo Controlled Study"
Brief Title: Intranasal Cooling for Symptomatic Relief of Migraine
Acronym: COOLHEAD2
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to insolvency of sponsor
Sponsor: Cumbria Partnership NHS Foundation Trust (Other)
Collaborators: BeneChill, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 3414
Record Dates: First submitted 2015-01-22; First posted 2015-03-03 (Estimated); Last update posted 2017-02-03 (Estimated); Status verified 2017-02

CONDITIONS: Migraine Headache
Keywords: Migraine Headache; Cooling; Intranasal; Rhinochill
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active RhinoChill (Active Comparator): Following the initial 30 days (and minimum of 2 separate migraine attacks) of data collection the patient will be trained in the use and self administration of the RhinoChill device.
  At the onset of an acute migraine, the patient will insert the RhinoChill Migraine Intranasal catheters and commence a 10 minute treatment on the Low Flow setting of the device.
  During this time the patient will complete the basic data record sheets to document current symptoms and changes in severity throughout the period of treatment and then at specific time points thereafter.
  The patient remains in the trial until two separate migraines have been treated.
  Interventions: Device: Active RhinoChill
- Placebo RhinoChill (Placebo Comparator): The same procedure will be followed for the placebo comparator as in the active comparator. The RhinoChill device looks identical and functions in a very similar way to the active device however through some minor design changes the device has been altered to provide a sufficient placebo treatment.
  At the onset of an acute migraine headache the patient will insert the RhinoChill Migraine Intranasal catheters and the 10 minute treatment is commenced on Low Flow.
  During this time the patient will complete the basic data record sheets to document current symptoms and changes in severity throughout the period of treatment and then at specific time points thereafter.
  The patient remains in the trial until two separate migraines have been treated.
  Interventions: Device: Placebo RhinoChill

INTERVENTIONS:
Device: Active RhinoChill — The device is intended for use for the reduction of temperature via the nasal cavity.
  The RhinoChill® System is a British Standards Institution Kite-Marked device that is currently commercially available in Europe. The RhinoChill® device is intended for temperature reduction in patients via the nasal cavity.
  Other Names: RhinoChill
  Arms: Active RhinoChill
Device: Placebo RhinoChill — The placebo RhinoChill device looks and functions in an identical way to the active RhinoChill. All components are used, however through some minor changes in the design of the device it now provides a sufficient placebo treatment to the patient.
  Other Names: RhinoChill
  Arms: Placebo RhinoChill

SUMMARY:
This study will be a randomised placebo controlled trial examining the effectiveness of using an intranasal cooling device (the RhinoChill) in providing relief of pain and symptoms of acute migraine. It will involve using two nasal catheters to cool the nasal cavity which provides localised cooling of the local nasal tissue and the blood vessels which supply blood to the brain. This cooling effect will cause the blood vessels to constrict as well as stimulating special cold receptors that are thought to be involved in the relief of migraine, thereby providing both pain and associated symptomatic relief. Ninety patients will be randomised in a 1:1 fashion, clustered to three different recruitment sites. The patients will have a 30 day period of data collection for their current migraine frequency, treatment and response to medication (with a minimum of 2 migraine attacks recorded) before starting the treatment phase with the RhinoChill Device. Treatment will be for 2 migraine attacks. Only a single treatment is allowed for the first attack, but on the second attack the patient may deliver 2 treatments with a gap of at least 2 hours between treatments.

DETAILED DESCRIPTION:
This study is a multi centre, double blinded, randomized, prospective, parallel placebo controlled trial for demonstrating the effectiveness of the RhinoChill System for the symptomatic relief of migraine headache.

The specific study design consists of:

* Participant identification from neurology clinic records and gaining initial consent to transfer contact details to the trial team.
* Telephone contact or direct clinic contact with potential participants to describe the COOLHEAD 2 trial and to seek expressions of interest.
* Initial meetings with potential participants and discussion of trial, provision of patient information leaflets. Informed Consent taking.
* Initial 30 day prospective data collection period (minimum of 2 migraine attacks, longer period if needed)
* Randomisation to either placebo or active RhinoChill
* Device Delivery and training session for the use of the RhinoChill device, self administration, and record keeping.
* Treatment period for the treatment of 2 separate migraines with the RhinoChill.

During an initial screening visit or phonecall, the trial will be discussed with the potential participant and the inclusion/exclusion checklist will be completed.

If the patient meets all inclusion criteria and none of the exclusion criteria, they will be asked for permission to pass on contact details to a member of the trial team for further contact.

Arrangements will then be made for a meeting with the patient either at the clinic or in their own home to further discuss the trial and to consider enrolling into the study. At this time, they will be provided with a patient information sheet and will be shown the RhinoChill device. The patient will be given the opportunity to fully consider all aspects of participation in this trial and to discuss it with family members if they so wish before being being consented into the trial by a member of the study team.

At the time of consent, the researcher will also collect data for the baseline CRF and provide initial instruction on completion of the first stage data collection forms (further described below)

At the baseline visit, the patient will first be given the opportunity to ask any questions they may have about the research. A member of the research team will take informed consent and gain signatures on the consent form. Baseline data will then be collected, including history of migraine headache, frequency, severity of symptoms, medication and therapies currently ongoing or taken in the past. Base line vital signs will also be recorded at this time. Once completed, a short training session on completion of the prospective data collection forms for phase 1 of the trial will given and use of the supplied blood pressure machine and pulse oxymeter machine. Once the baseline visit has been completed the patient will begin a 30 day period of self data collection based on their migraine experience during that time frame and using data capture forms provided by the research nurse (a minimum of 2 migraine attacks are required, therefore if 2 have not occurred during the 30 days, further time will be given to allow the second migraine to occur).

If a patient has not had a single migraine in the first 30 days, then they will not be able to continue to the treatment phase as they have not met the inclusion criteria of at least 1 migraine per month. Following the conclusion to this initial period, the treatment phase will then begin.

After the end of the prospective data collection period, the patient will be randomised to either active treatment or placebo treatment. Randomisation will be provided by sealed envelopes held by E&E CRO services (Vienna) who are also acting as independent monitors of the trial. Randomisation was performed via the online system www.sealedenvelope.com.

Training will be undertaken to ensure that the patient is fully competent and safe in the use of the RhinoChill intranasal cooling device.

The patient will be instructed on:

* Preparation of the device
* Insertion of the nasal catheter
* Selecting correct flow rate
* Positioning during treatment
* Cleaning and storage of the nasal catheters
* Trial documentation
* 24 hour contact numbers for additional supplies, troubleshooting and practical support.

The patient will also be left with a reference booklet for issues around the trial and the practical use of the RhinoChill device.

At the onset of migraine headache (or as soon as possible thereafter), the patient will start to complete the 'Treatment' CRF.

Each step of the treatment procedure is to be completed in order and as described to the patient. Patients are instructed that there is no scope for any alteration in the treatment order or requirements of the trial unless a safety issue becomes evident. If a patient does deviate from the standard procedures as outlined below, they are required to contact the 24 hour COOLHEAD 2 mobile phone to report the incident so that it can be reviewed and logged as a protocol deviation and reviewed by the site/principal investigator at the earliest opportunity. The RhinoChill device is then prepared for use and treatment can be administered.

The RhinoChill Migraine Intranasal catheters are then inserted and the 10 minute treatment is commenced on Low Flow. following these steps for each individual treatment:

It is recognised that participants in this study will already be taking medication for their migraine headache. Normal prophylaxis will be allowed as part of the trial and will be recorded in the initial screening interview. No change in prophylaxis is allowed within three months of the start of the trial or while the patient is participating in the trial.

However, acute treatments such as triptans are allowed to be taken but must be withheld until at least two hours following completion of treatment with the RhinoChill to allow assessment of the intervention. Any rescue medication taken after this point will be recorded in the associated trial documentation. A full medication history along with other therapies (including alternative therapies) will also be recorded.

No new treatment or therapy will start while the participant is enrolled in this trial.

ELIGIBILITY:
Inclusion Criteria:

* 18 Years or over and ≤70 years of age.
* Migraine diagnosis of at least 1 year.
* Migraine attacks between 1 and 15 per month.
* Onset of first migraine < 50 years of age.
* Migraine prophylaxis medication unchanged for 3 months prior to enrollment
* Meets International Classification for Headache Disorders (2nd Edition) criteria for diagnosis of Episodic Migraine with or without aura
* Able to attend and understand a short training session on the practical use of the RhinoChill device and agrees to only use the device as instructed and as laid out in the official instructions for use.

Exclusion Criteria:

* < 18 and >70 years of age
* Known oxygen dependency to maintain SaO2 >95%
* Diagnosed Hypertensive and currently uncontrolled with Systolic BP > 140mmHg and Diastolic BP > 90mmHg on baseline assessment.
* Marked nasal septal deviation, recurrent epistaxis or chronic Rhino-Sinusitis
* Intranasal obstruction preventing full insertion of nasal catheter
* Known acute base of skull fracture or facial trauma
* Concurrent sinus/intranasal surgery
* Diagnosed with thromobocytopenia.
* Previous Stroke or Myocardial Infarction
* Unable to fully understand the consent process and provide informed consent due to either language barriers or mental capacity
* Previously enrolled into the COOLHEAD 1 trial
* No recorded migraine following initial 30 day data collection period

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Pain free at two hours following treatment | Two hours following treatment
  Percentage of patients who are pain free two hours following treatment

SECONDARY OUTCOMES:
Percentage of patients pain free | 10 mins, 1 hour, 2 hours, 24 hours
  Percentage of patients scoring a pain intensity score of None
Headache response | 10 mins, 1 hour, 24 hours
  Headache response - Improvement of pain from Severe/Moderate to mild/none immediately following treatment and at one hour and 24 hours following treatment.
Pain response | 10 mins, 1 hour, 2 hours, 24 hours
  Change in pain score (Visual Analogue Score of 0-10) immediately following treatment and at one hour, 2 hours and 24 hours following treatment.
Relapse Incidence | Between 2 and 48 hours after the intervention
  Relapse Incidence - Frequency of headache return between 2 and 48 hours after the intervention
Sustained Pain Freedom | Between 1 and 24 hours after the intervention
  Pain free at 2 hours with no use of rescue medication or relapse within the subsequent 46 hours
Total Migraine Freedom | Between 1 and 24 hours after the intervention
  Absence of pain, nausea, photophobia and phonophobia at 2 hours
Change in Headache Intensity during treatment. | 5 mins and 10 mins
  Change in Headache Intensity during treatment.
Change in Headache Intensity 2 hours following treatment | 2 hours following treatment.
  Change in Headache Intensity 2 hours following treatment
Time to meaningful relief | Between 10 mins and 24 hours after the intervention
  Time to meaningful relief. Time to meaningful relief Time to freedom from pain
Time to freedom from pain | Between 10 mins and 24 hours after the intervention
  Time to freedom from pain Time to meaningful relief Time to freedom from pain
Percentage of patients taking rescue medication at 2 hours after treatment | 2 hours after treatment
  Percentage of patients taking rescue medication at 2 hours after treatment
Global Impression of Change | to be completed at the end of trial period, an average of 8-10 weeks
  Global Impression of Change
Global impact on disability. | to be completed at the end of trial period, an average of 12 weeks
  Global impact on disability. Global impact on disability and Quality of life
Global impact on quality of life | to be completed at the end of trial period, an average of 12 weeks
  Global impact on quality of life Global impact on disability and Quality of life
Impact on migraine associated symptoms | To be measured at 10 mins, 1 hour, 2 hours, 24 hours
  Impact on migraine associated symptoms:
  Nausea Photophobia Phonophobia
Migraine pain scores, pre intervention data collection period versus treatment with the intervention. | to be completed at the end of trial period, an average of 12 weeks
  Migraine pain score, pre intervention data collection period versus treatment with the intervention.
Comparison of symptoms scores between pre intervention data collection period and treatment with the intervention. | to be completed at the end of trial period, an average of 12 weeks
  Comparison of symptoms scores between pre intervention data collection period and treatment with the intervention.
  * Headache severity Severe/moderate - mild/none
  * VAS score (0-10 pain scale & Symptom severity)
Adverse events | From day one of the intervention period until 48 hours post 2nd trial treatment
  Adverse events noted throughout the treatment phase and during follow up

CONTACTS AND LOCATIONS:
Overall Officials: Jitka Vanderpol, MD FRCP, Principal Investigator — Cumbria Partnership NHS Foundation Trust
Locations (3):
- United Kingdom (3):
  - Neurosciences department, Penrith Hospital, Cumbria Partnership NHS Foundation Trust, Penrith, Cumbria
  - CITY HOSPITALS SUNDERLAND NHS FOUNDATION TRUST, 11 Norfolk Street, Sunderland SR1 1EA, Sunderland, Tyne and Wear
  - The James Cook University Hospital, South Tees Hospitals NHS Foundation Trust, Middlesbrough

REFERENCES:
- [Background] Zanchin G, Maggioni F, Granella F, Rossi P, Falco L, Manzoni GC. Self-administered pain-relieving manoeuvres in primary headaches. Cephalalgia. 2001 Sep;21(7):718-26. doi: 10.1046/j.1468-2982.2001.00199.x. PMID 11594999
- [Background] Ucler S, Coskun O, Inan LE, Kanatli Y. Cold Therapy in Migraine Patients: Open-label, Non-controlled, Pilot Study. Evid Based Complement Alternat Med. 2006 Dec;3(4):489-93. doi: 10.1093/ecam/nel035. Epub 2006 Jun 15. PMID 17173113
- [Background] Diamond S, Freitag FG. Cold as an adjunctive therapy for headache. Postgrad Med. 1986 Jan;79(1):305-9. doi: 10.1080/00325481.1986.11699255. PMID 3941818
- [Background] Robbins LD. Cryotherapy for headache. Headache. 1989 Oct;29(9):598-600. doi: 10.1111/j.1526-4610.1989.hed2909598.x. PMID 2584002
- [Background] Lance JW. The controlled application of cold and heat by a new device (Migra-lief apparatus) in the treatment of headache. Headache. 1988 Aug;28(7):458-61. doi: 10.1111/j.1526-4610.1988.hed2807458.x. No abstract available. PMID 3243707
- [Background] Friedman MH, Peterson SJ, Behar CF, Zaidi Z. Intraoral chilling versus oral sumatriptan for acute migraine. Heart Dis. 2001 Nov-Dec;3(6):357-61. doi: 10.1097/00132580-200111000-00003. PMID 11975819
- [Background] Sprouse-Blum AS, Gabriel AK, Brown JP, Yee MH. Randomized controlled trial: targeted neck cooling in the treatment of the migraine patient. Hawaii J Med Public Health. 2013 Jul;72(7):237-41. PMID 23901394
- [Background] ABRAMSON DI. PHYSIOLOGIC BASIS FOR THE USE OF PHYSICAL AGENTS IN PERIPHERAL VASCULAR DISORDERS. Arch Phys Med Rehabil. 1965 Mar;46:216-44. No abstract available. PMID 14271050
- [Background] Swenson C, Sward L, Karlsson J. Cryotherapy in sports medicine. Scand J Med Sci Sports. 1996 Aug;6(4):193-200. doi: 10.1111/j.1600-0838.1996.tb00090.x. PMID 8896090
- [Background] Dolan MG, Thornton RM, Fish DR, Mendel FC. Effects of cold water immersion on edema formation after blunt injury to the hind limbs of rats. J Athl Train. 1997 Jul;32(3):233-7. PMID 16558455
- [Background] Deal DN, Tipton J, Rosencrance E, Curl WW, Smith TL. Ice reduces edema. A study of microvascular permeability in rats. J Bone Joint Surg Am. 2002 Sep;84(9):1573-8. PMID 12208913
- [Background] De Jong RH, Hershey WN, Wagman IH. Nerve conduction velocity during hypothermia in man. Anesthesiology. 1966 Nov-Dec;27(6):805-10. doi: 10.1097/00000542-196611000-00013. No abstract available. PMID 5924554
- [Background] Merrick MA. Secondary injury after musculoskeletal trauma: a review and update. J Athl Train. 2002 Apr;37(2):209-17. PMID 16558673
- [Background] Zachariassen KE. Hypothermia and cellular physiology. Arctic Med Res. 1991;50 Suppl 6:13-7. PMID 1811567
- [Background] Numazaki M, Tominaga M. Nociception and TRP Channels. Curr Drug Targets CNS Neurol Disord. 2004 Dec;3(6):479-85. doi: 10.2174/1568007043336789. PMID 15578965
- [Background] Zenker W, Kubik S. Brain cooling in humans--anatomical considerations. Anat Embryol (Berl). 1996 Jan;193(1):1-13. doi: 10.1007/BF00186829. PMID 8838492
- [Background] Van den Brande P, De Coninck A, Lievens P. Skin microcirculation responses to severe local cooling. Int J Microcirc Clin Exp. 1997 Mar-Apr;17(2):55-60. doi: 10.1159/000179207. PMID 9253681
- [Background] Boller M, Lampe JW, Katz JM, Barbut D, Becker LB. Feasibility of intra-arrest hypothermia induction: A novel nasopharyngeal approach achieves preferential brain cooling. Resuscitation. 2010 Aug;81(8):1025-30. doi: 10.1016/j.resuscitation.2010.04.005. Epub 2010 Jun 9. PMID 20538402
- [Background] Wang H, Barbut D, Tsai MS, Sun S, Weil MH, Tang W. Intra-arrest selective brain cooling improves success of resuscitation in a porcine model of prolonged cardiac arrest. Resuscitation. 2010 May;81(5):617-21. doi: 10.1016/j.resuscitation.2010.01.027. Epub 2010 Mar 6. PMID 20207471
- [Background] Yu T, Barbut D, Ristagno G, Cho JH, Sun S, Li Y, Weil MH, Tang W. Survival and neurological outcomes after nasopharyngeal cooling or peripheral vein cold saline infusion initiated during cardiopulmonary resuscitation in a porcine model of prolonged cardiac arrest. Crit Care Med. 2010 Mar;38(3):916-21. doi: 10.1097/CCM.0b013e3181cd1291. PMID 20081534
- [Background] Tsai MS, Barbut D, Tang W, Wang H, Guan J, Wang T, Sun S, Inderbitzen B, Weil MH. Rapid head cooling initiated coincident with cardiopulmonary resuscitation improves success of defibrillation and post-resuscitation myocardial function in a porcine model of prolonged cardiac arrest. J Am Coll Cardiol. 2008 May 20;51(20):1988-90. doi: 10.1016/j.jacc.2007.12.057. No abstract available. PMID 18482670
- [Background] Guan J, Barbut D, Wang H, Li Y, Tsai MS, Sun S, Inderbitzen B, Weil MH, Tang W. A comparison between head cooling begun during cardiopulmonary resuscitation and surface cooling after resuscitation in a pig model of cardiac arrest. Crit Care Med. 2008 Nov;36(11 Suppl):S428-33. doi: 10.1097/ccm.0b013e31818a8876. PMID 20449906
- [Background] Abou-Chebl A, Sung G, Barbut D, Torbey M. Local brain temperature reduction through intranasal cooling with the RhinoChill device: preliminary safety data in brain-injured patients. Stroke. 2011 Aug;42(8):2164-9. doi: 10.1161/STROKEAHA.110.613000. Epub 2011 Jun 16. PMID 21680904
- [Background] Busch HJ, Eichwede F, Fodisch M, Taccone FS, Wobker G, Schwab T, Hopf HB, Tonner P, Hachimi-Idrissi S, Martens P, Fritz H, Bode Ch, Vincent JL, Inderbitzen B, Barbut D, Sterz F, Janata A. Safety and feasibility of nasopharyngeal evaporative cooling in the emergency department setting in survivors of cardiac arrest. Resuscitation. 2010 Aug;81(8):943-9. doi: 10.1016/j.resuscitation.2010.04.027. Epub 2010 Jun 2. PMID 20627524
- [Background] Castren M, Nordberg P, Svensson L, Taccone F, Vincent JL, Desruelles D, Eichwede F, Mols P, Schwab T, Vergnion M, Storm C, Pesenti A, Pachl J, Guerisse F, Elste T, Roessler M, Fritz H, Durnez P, Busch HJ, Inderbitzen B, Barbut D. Intra-arrest transnasal evaporative cooling: a randomized, prehospital, multicenter study (PRINCE: Pre-ROSC IntraNasal Cooling Effectiveness). Circulation. 2010 Aug 17;122(7):729-36. doi: 10.1161/CIRCULATIONAHA.109.931691. Epub 2010 Aug 2. PMID 20679548
- [Background] Tfelt-Hansen P, Pascual J, Ramadan N, Dahlof C, D'Amico D, Diener HC, Hansen JM, Lanteri-Minet M, Loder E, McCrory D, Plancade S, Schwedt T; International Headache Society Clinical Trials Subcommittee. Guidelines for controlled trials of drugs in migraine: third edition. A guide for investigators. Cephalalgia. 2012 Jan;32(1):6-38. doi: 10.1177/0333102411417901. No abstract available. PMID 22384463